CLINICAL TRIAL: NCT06812039
Title: HAIC Combined with Donafenib and Sintilimab As Perioperative Treatment for Resectable Hepatocellular Carcinoma Patients At High Risk of Recurrence: a Prospective, Multicenter, Randomized Phase II Study
Brief Title: HAIC Combined with Donafenib and Sintilimab As Perioperative Treatment for Resectable Hepatocellular Carcinoma Patients At High Risk of Recurrence
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Lu Wang, MD, PhD, Professor, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2412311-5
Record Dates: First submitted 2025-01-19; First posted 2025-02-06 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Hepato Cellular Carcinoma (HCC)
MeSH Terms: interventions — sintilimab; donafenib; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group A (Experimental): HAIC combined with sintilimab and donafenib
  Interventions: Drug: HAIC combined with sintilimab and donafenib
- Group B (Experimental): Sintilimab and Donafenib
  Interventions: Drug: Sintilimab and Donafenib
- Group C (Active Comparator): Direct surgery
  Interventions: Procedure: Surgery

INTERVENTIONS:
Drug: HAIC combined with sintilimab and donafenib — HAIC: Two cycles, Q3W. The chemotherapy regimen consists of oxaliplatin 85 mg/m² over 2 hours and raltitrexed 2 mg/m² over 1 hour.
  Donafenib: Treatment should begin the day after the completion of the first HAIC, with an initial dose of 0.1g bid p.o.. The investigator may increase the dose to 0.2g bid depending on the patient's condition.
  Sintilimab: Administration may begin after the first HAIC, 200 mg iv Q3W. After surgery, continued sintilimab and donafenib for 6 cycles.
  Arms: Group A
Drug: Sintilimab and Donafenib — Donafenib: an initial dose of 0.1g bid p.o. The investigator may increase the dose to 0.2g bid depending on the patient's condition. Sintilimab: 200 mg iv Q3W. After surgery, continued sintilimab and donafenib for 6 cycles.
  Arms: Group B
Procedure: Surgery — After surgery, received sintilimab and donafenib for 6 cycles.
  Arms: Group C

SUMMARY:
This study will evaluate the efficacy and safety of therapy perioperative treatment with HAIC combined with donafenib and sintilimab (group A)/ donafenib combined with sintilimab (group B) compared with direct surgery (group C) in resectable HCC patients who are at high risk for disease recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary enrollment with written informed consent obtained
* Age 18 to 75 years (inclusive), regardless of gender
* Histologically or pathologically confirmed previously untreated hepatocellular carcinoma (HCC) or clinically diagnosed previously untreated HCC according to the AASLD guidelines.
* Initial resectable status as assessed by the investigator (expected to achieve R0 resection, sufficient liver remnant volume, and Child-Pugh class A, as per the "Chinese Expert Consensus on Neoadjuvant Therapy for Liver Cancer (2023 Edition)").
* At least one measurable lesion according to mRECIST criteria.
* Tumor burden meets one of the following conditions:

  1. A single tumor with a diameter > 5 cm;
  2. Multiple tumors with the largest tumor diameter > 3 cm, with < 5 tumors in total;
  3. Presence of portal vein tumor thrombus (Vp1-Vp2).
* Liver function: Child-Pugh score of 5-6.
* ECOG 0-1
* Life expectancy of at least 3 months.
* Women of childbearing potential (defined as not postmenopausal or surgically sterilized) must have a negative serum pregnancy test within 7 days prior to the study drug administration.
* Both women and men of childbearing potential must use reliable contraception during the study and for 60 days following the last dose of the study drug.
* For HBV-infected patients: If HBV-DNA is ≥ 10⁴ copies/ml within 14 days prior to enrollment, antiviral therapy (preferably entecavir) must be initiated to reduce HBV-DNA to < 10⁴ copies/ml before entering the study. Antiviral therapy should continue, with regular monitoring of liver function and HBV-DNA levels.
* Adequate organ function.

Exclusion Criteria:

* Patients with distant metastasis.
* Patients with portal vein tumor thrombosis (Vp3-Vp4).
* History of any other malignant tumor within the past 5 years, unless the patient has received potentially curative treatment and there is no evidence of recurrence in the past 5 years. This 5-year time requirement does not apply to patients who have successfully undergone resection for basal cell carcinoma of the skin, squamous cell carcinoma of the skin, superficial bladder cancer, cervical carcinoma in situ, or other carcinoma in situ.
* History or current presence of congenital or acquired immunodeficiency diseases.
* Active or previously documented autoimmune diseases or inflammatory disorders (including but not limited to: autoimmune hepatitis, interstitial pneumonia, inflammatory bowel disease, systemic lupus erythematosus, vasculitis, uveitis, pituitary inflammation, hyperthyroidism or hypothyroidism, asthma requiring bronchodilators for treatment, etc.). Patients with vitiligo or asthma fully resolved in childhood and not requiring intervention as adults may be included.
* History of severe psychiatric disorders.
* Conditions affecting the absorption, distribution, metabolism, or elimination of the study drugs (e.g., severe vomiting, chronic diarrhea, bowel obstruction, malabsorption, etc.).
* Major surgery within 4 weeks prior to enrollment (as defined by the investigator).
* History of allogeneic stem cell or solid organ transplantation (except for corneal transplantation).
* Received other systemic antitumor therapies (including traditional Chinese medicine with antitumor indications) within 2 weeks or 5 half-lives (whichever is longer) prior to study drug administration, or unresolved adverse events related to prior treatments that have not recovered to ≤ CTCAE Grade 1.
* Use of systemic immunosuppressive drugs within 2 weeks prior to enrollment, or anticipated need for systemic immunosuppressive therapy during the study.
* Concurrent use of drugs that may prolong the QTc interval and/or induce Tdp, or drugs affecting drug metabolism.
* Known or suspected allergy to donafenib, recombinant humanized PD-1 monoclonal antibodies, or similar agents, or a history of hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins, or to excipients of the study drugs.
* Uncontrolled hepatic encephalopathy, hepatorenal syndrome, ascites, pleural effusion, or pericardial effusion.
* Active bleeding or coagulation disorders, bleeding tendencies, or ongoing treatment with thrombolytics, anticoagulants, or antiplatelet therapy.
* History of gastrointestinal bleeding or clear gastrointestinal bleeding tendencies within the past 6 months (e.g., known active ulcerative lesions, positive stool occult blood with ≥2+ results, requiring endoscopy if stool occult blood remains positive), or other conditions that may lead to gastrointestinal bleeding as determined by the investigator (e.g., severe esophageal/gastric varices).
* History of gastrointestinal perforation, abdominal fistulas, or intra-abdominal abscesses within the past 6 months.
* History of thrombosis or thromboembolic events (e.g., stroke, transient ischemic attack, deep vein thrombosis, pulmonary embolism) within the past 6 months.
* Significant cardiovascular disease, including but not limited to: acute myocardial infarction, severe/uncontrolled angina, coronary artery bypass grafting within the past 6 months; congestive heart failure (NYHA class >2); poorly controlled arrhythmias requiring pacemaker treatment; drug-resistant hypertension (systolic blood pressure ≥140 mmHg and/or diastolic blood pressure ≥90 mmHg).
* Active infection.
* Other significant clinical or laboratory abnormalities that may affect safety evaluation, such as uncontrolled diabetes, chronic kidney disease, grade 2 or higher peripheral neuropathy (CTCAE v5.0), thyroid dysfunction, etc.
* Use of live attenuated vaccines within 4 weeks prior to enrollment or during the study.
* Pregnant or breastfeeding women, or women or men of childbearing potential unwilling or unable to use effective contraception.
* History of alcohol, drug, or substance abuse within the past 6 months.
* Participation in any other clinical trial involving investigational drugs or medical devices within 4 weeks prior to enrollment.
* Inability to comply with the study protocol for treatment or follow-up visits.
* Any other conditions that, in the opinion of the investigator, would preclude participation in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
1-yr RFS rate | 24 months
  the proportion of patients who have not experienced recurrence or death from any cause at 12 months after hepatectomy.

SECONDARY OUTCOMES:
MPR rate | Up to approximately 12 weeks
  The percentage of patients with 70%-99% tumor necrosis found during surgery after neoadjuvant therapy
pCR rate | Up to approximately 12 weeks
  the percentage of participants having a pathCR
ORR | Up to approximately 12 weeks
  The percentage of subjects in the overall population who achieved CR or PR according to the mRECIST criteria
RFS | Up to approximately 2 years
  RFS is defined as the time from liver resection to the first documented occurrence of intrahepatic or extrahepatic HCC, or death from any cause (whichever occurs first).
PFS | Up to approximately 2 years
  PFS is defined as the time from randomization to the first documented occurrence of intrahepatic or extrahepatic HCC, or death from any cause (whichever occurs first).
OS | Up to approximately 3 years
  OS is defined as the time from randomization to death from any cause.
TTR | Up to approximately 2 years
  TTR is defined as the time from liver resection to the first documented occurrence of intrahepatic or extrahepatic HCC.

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - TianJin Medical University Cancer Institute & Hospital, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: No